CLINICAL TRIAL: NCT05797727
Title: LIFECHAMPS: A Collective Intelligence Platform to Support Cancer Champions Real-Life Pilot
Brief Title: Real-Life Pilot Feasibility Study (LC_RLP)
Acronym: LC_RLP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: University of Glasgow (Other); Region Stockholm (Other Government); Hospital Universitario La Fe (Other)
Responsible Party: Principal Investigator, Panos Bamidis, Professor, Aristotle University Of Thessaloniki
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 875329B
Record Dates: First submitted 2023-03-22; First posted 2023-04-04 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer; Prostate Cancer
Keywords: Cancer; mHealth App; Ambient Sensors; Wearables; Smartwatch; Smart scale; Analytics Engine
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms; Neoplasms

STUDY DESIGN:
Intervention Model Description: Parallel: Clinical trials with a two arms: A prospective, pre-post design will be employed, whereby the LifeChamps platform will be deployed for a total of 3 months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LifeChamps Platform (Experimental): Participants will be asked to use the LifeChamps platform and will be provided with the study equipment.
  Interventions: Device: LifeChamps Platform
- LifeChamps Platform HCP (Experimental): Participating Healthcare professionals will be asked to use the LifeChamps Dashboard
  Interventions: Device: LifeChamps Platform HCP

INTERVENTIONS:
Device: LifeChamps Platform HCP — Healthcare professionals that will participate in the study will be introduced will have access to the LifeChamps Dashboard, which will display the data monitored from the patients, thus potentially facilitating patients' follow-up between clinical consultations. The LC Dashboard will provide pseudonymised information regarding the patients' physical activity and PROMs for the purpose of the pilot feasibility trial. They will not be able to view real time processed information, such as risk of frailty, QoL, risk of dependency and psychological condition, from the LIFECHAMPS analytics engine. They will be shown the anonymised outputs of the engine per patient and asked their opinions on the usability, acceptability and on whether such information would have helped better manage their patients' supportive care.
  Arms: LifeChamps Platform HCP
Device: LifeChamps Platform — Participants will be asked to provide 5 endpoints (PROMS) and will be provided with the study equipment, i.e., a mobile app, smartwatch, smart scale, location home sensor, a smart plug, and a micro-computer, with which they will need to interact with the devices for three months. Specifically, participants should wear the activity tracker wristband (Fitbit Charge 4) as much as possible. Additionally, participants should use the smart scale to weigh themselves and the mobile app to fill in selected PROMs monthly, while the ambient home sensors will be passively collecting information about their everyday living during these three months. At the end of the 3 month period, the participants will return the devices and will be asked to provide the 5 endpoints and their opinions regarding the usability and acceptability of the platform using structured questionnaires
  Arms: LifeChamps Platform

SUMMARY:
The LifeChamps Real-Life pilot's objective is to ascertain the feasibility of the use of the LifeChamps solution, previously developed in another clinical trial, in a real-world environment. This solution integrates a health advisory system, and technical intelligence, based on behavioural science, to provide personalized recommendations to follow a healthier lifestyle, to act as a nutrition and physical activity coach, and to guide on social inclusion, among other issues, with the aim of increasing the quality of life. This study is conducted to investigate the feasibility of such an undertaking, assess the clinical impact it may have, as well as evaluate the applicability, usability, and effectiveness of the solution.

DETAILED DESCRIPTION:
"The LifeChamps project (https://lifechamps.eu/) is creating a digital platform to support clinical teams to provide more integrated follow-up care to older patients with cancer. The digital platform will integrate data coming directly from the patient (patient-reported outcomes and sensor data from wearable devices), from the home environment (home sensors, weight scales), and from the clinical environment (data routinely collected via the Electronic Health Record). The digital platform will use big data analytics (machine learning) to process all data as part of predictive clinical algorithms for frailty and quality of life for older patients with cancer. Development of each clinical algorithm requires that the prototype model (or analytics engine) is trained using abundant real-world data to help consolidate the predictive ability and validity of the algorithms before the algorithms are deployed in a larger scale feasibility trial.

A pre-post design will be employed, whereby the LifeChamps platform will be deployed for a total of 3 months.

The main research questions of the study are:

1. Is patient recruitment possible in terms of numbers and rates within the recruitment period?
2. Is participant retention in the study possible in terms of numbers and rates?
3. Do participants adhere to the protocol?
4. What are the views/experiences of study participants (patients and healthcare professionals) using the Lifechamps solution (mHealth app and dashboard respectively)?
5. What is the adherence with the usage of the different digital health patients' tools (e.g., usage of mHealth app, smartwatch, smart weight scale)?

Healthcare professionals related to oncology (oncologists, nurses etc.) will also be recruited to use the LifeChamps dashboard and evaluate its usefulness, usability and acceptability. They will have access to and asked to use the LC Dashboard. The LC Dashboard will provide pseudonymised information regarding the patients' physical activity and PROMs for the purpose of the pilot feasibility trial. They will not be able to view real time processed information. After the patients have exited the study, the HCPs will be shown the anonymised outputs of the engine per patient and asked their opinions.

Older patients with a cancer diagnosis will be the target population for this study. Target number of participants is 200. Each study participant will be involved in the study for 3 months in total. A 4-month recruitment period will be allowed, bringing the total study duration to 7 months (from first patient being enrolled until last patient finishing data collection).

After written informed consent has been provided, the mini-COG will be used to evaluate study participants' cognitive function and impairment at baseline. The mini-COG consists of a 3-word recall and a clock-drawing test, and can be completed within 5 minutes. A score of less than 3/5 indicates the need to refer the patient for full cognitive assessment. Study endpoints will be collected at this point.

The researcher will also arrange for study participants to receive study equipment, i.e. home sensors, wearable activity sensors, smart weight scale, and mobile app. The researcher will arrange a suitable time for a home visit to install the home sensors and test functionality. The researcher will demonstrate use of study equipment to the participant, and reiterate that support with use of the technology will be available.

Data collection will involve a variety of sources, including the patient (patient-reported outcomes and sensor data from wearable devices), the home environment (home sensors, weight scales), and the clinical site (data routinely collected via the Electronic Health Record).

The following technology will be used:

Mobile devices:

Activity tracker wristband (FitBit charge 4). It will be used to passively monitor and collect data on heart rate, heart rate variability, steps, activity tracking, sleep monitoring, breathing rate, skin temperature and SpO2.

mHealth app (SALUMEDIA). It will be used to enable collection of patient-reported outcome measures (PROMs) and to forward this information along with the data gathered by the activity tracker and the smart scale to the Raspberry Pi Kit at home.

At home sensors / devices:

LOCS Home sensors: They will be used to monitor participants' daily activities e.g., to track ambulation and functioning. Study participants will be provided with 4 motion sensors, 1 door contact sensor, 2 corridor sensors, and a tag device.

Smart Scale (Withings Body+): It will be used to measure weekly body weight, body composition and body mass index.

Raspberry Pi (RPI) kit: As an edge gateway, RPI is hosting LOCS gateway, Movesense Gateway and data ingestion service. RPI will enable data collection and edge analytics and transfer of data to the LIFECHAMPS platform.

Smart plug: It will be used to collect data about use home appliances and thereby data about active daily living.

Selected study participant clinical and demographic data from the local EHRs will be collected and loaded onto the LifeChamps analytics engine. The data will be loaded by technical partners via the LifeChamps dashboard for processing and analysis. Data regarding recruitment rate (patients consenting / patients approached), participant retention in the study, reasons for study discontinuation (if offered), participant adherence with technology, issues with technology and need for troubleshooting will be recorded. These data will (a) be recorded by local researchers using bespoke 'recording logs' in the form of an Excel spreadsheet, and (b) remotely monitored and logged by technical partners involved in the distribution / management of the technology to be used in the trial as described above."

ELIGIBILITY:
Inclusion Criteria:

* Breast or prostate cancer.
* Diagnosed with early stage (I-III) cancer (breast, prostate) and living beyond initial cancer treatment (curative/incurable).
* Diagnosed with advanced or metastatic disease with life expectancy >12 months.
* At least 1 month after a) local treatment with curative intent (surgery, radiotherapy) or b) initiation of systemic treatment (hormone treatment, CDK4/6 or new generation antiandrogens).
* Absence of diagnosed secondary malignancy.
* Deemed by a member of the multidisciplinary team as physically and psychologically fit to participate in the study.
* Able to read, write and understand the respective local language (greek).
* Achieve a score of above 2 on the Mini-Cog during the screening process.
* Able to bring and use own Android version 10 (or above) device during the study.
* Domestic 24/7 internet access via wi-fi and/or 4G mobile data (will be provided if unavailable).

Exclusion Criteria:

* Currently receiving chemotherapy.
* Terminal cancer stage on palliative care.
* Survival prognosis of <18 months from the time of recruitment.
* Unwilling to provide written informed consent.
* Presence of internal medical device (e.g. pacemaker etc.)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 121 (Actual)
Dates: Start 2023-01-15 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-06 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | 7 months
  This outcome will be calculated by dividing the number of participants consented over the number of approached participants. It is a ratio between 0 and 1, with 1 being the best outcome.
Participant retention rate | 7 months
  This outcome will be calculated by dividing the number of participants that finished the study over the number of participants that entered the study. It is a ratio between 0 and 1, with 1 being the best outcome.
Technology Adherence rate | 7 months
  This outcome will be calculated by dividing the number of times the technology was used over the maximum times that technology can be used over the course of the study. It is a ratio between 0 and 1, with 1 being the best outcome.

SECONDARY OUTCOMES:
Quality of life Assessment | 3 months
  This outcome will be measured using the EQ-5D-5L questionnaire. It is using 5-Level Likert scale, with 0 being the best. Also, it includes a self-report of health status using a 0 to 100 scale, 100 being best.
Functional Assessment | 3 months
  This outcome will be measured using the Functional Assessment of Cancer Therapy - General - 7 Item Version (FACT-G7) Questionnaire. It uses a 5-Level Likert scale, 0 being the best.
Frailty | 3 months
  This outcome will be measured using the Tilburg Frailty Indicator. It uses Yes-No questions to calculate a score between 0 and 15, with 0 being the best.
Quality of Life Utility Measure | 3 months
  This outcome will be measured using the EORTC QUALITY OF LIFE UTILITY - CORE 10 DIMENSIONS (QLU-C10D) Questionnaire. It uses a 4-Level Likert scale, with 4 being the best.

OTHER OUTCOMES:
Perceived Acceptability | 3 months
  This outcome will be measured by structured custom made questionnaires, using a 5-level Likert Scale, with 5 representing high acceptance
Perceived Usability | 3 months
  This outcome will be measured by structured custom made questionnaires, using a 5-level Likert Scale, with 5 representing high usability

CONTACTS AND LOCATIONS:
Overall Officials: Panos D Bamidis, PhD, Principal Investigator — Aristotle University Of Thessaloniki
Locations (1):
- Laboratory of Medical Physics and Digital Innovation, AUTH, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: Yes
Data collected during the Real-Life pilot study, will be made available for sharing via open access repositories, according to the Final Version of the Data Managements Plan of the project.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be made available 5 years after the end of the study for indefinite period of time.
Access Criteria: Data will be made available only for non-commercial research purposes.